CLINICAL TRIAL: NCT00718354
Title: Randomized, Phase III-b, Multi-centre, Open-label, Parallel Study of Enoxaparin (Low Molecular Weight Heparin) Given Concomitantly With Chemotherapy vs Chemotherapy Alone in Patients With Inoperable Gastric and Gastro-oesophageal Cancer
Brief Title: Overall Survival of Inoperable Gastric/GastroOesophageal Cancer Subjects on Treating With LMWH + Chemotherapy(CT) vs Standard CT
Acronym: GASTRANOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thrombosis Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TRI0702
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Cancer; Gastroesophageal Cancer
Keywords: Bleeding events
MeSH Terms: conditions — Stomach Neoplasms | interventions — Enoxaparin; Epirubicin; Cisplatin; Capecitabine; XELOX; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator): Standard Chemotherapy (upto 6 cycles)
  Interventions: Drug: Standard Chemotherapy
- A (Experimental): Enoxaparin: 1 mg/kg once daily in addition to standard chemotherapy up to 6 months
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Once daily dose of 1mg/Kg of body weight for 6 months
  Arms: A
Drug: Standard Chemotherapy — Investigator's discretion
  Other Names: Some commonly prescribed Chemotherapy regimens in India are:; - Epirubicin + Cisplatin + Capecitabine; - Capecitabine + Oxaliplatin; - Docetaxil + Carboplatin; - Epirubicin + Cisplatin + Fluorouracil; - Docetaxil + Cisplatin with G/C/S/F support; - Epirubicin + Cisplatin + Flourouracil; - Docetaxil + Cisplatin + Flourouracil
  Arms: B

SUMMARY:
Due to evidence available both in terms of efficacy and safety of low molecular weight heparin, its use for the prevention of thromboembolic disease in cancer patients undergoing surgical intervention, and its extended use in higher doses for the prevention of recurrent thromboembolism in cancer patients with established thrombosis, with a view that the potential benefits for survival in cancer patients from low molecular weight heparin therapy comes because of a biological activity, the dose of 1mg/Kg (50% of the full treatment dose) for a period of 6 months coincident with 6 cycles of chemotherapy, has been chosen for this study.

DETAILED DESCRIPTION:
In the GASTRANOX study, patients will have inoperable (locally advanced) or metastatic newly diagnosed gastric or gastro oesophageal cancer. These patients carry a definite thrombosis risk. Patients will be scheduled to have at least 6 months of palliative chemotherapy. During this period symptomatic thromboembolism will be common but currently no routine prophylaxis is provided.

The dose of Enoxaparin to be evaluated in this study is 1mg/kg. This represents half of the full treatment dose. For an average weight individual this will represent between 60 and 70 mg a day of Enoxaparin. The prophylactic dose for high-risk surgical patients in the United States is 60mg total daily dosing of Enoxaparin per day. This high-risk dose has been shown to be safe and effective in preventing thromboembolic disease in high-risk populations such as those undergoing major elective orthopaedic surgery. An alternative for high-risk dose is 40mg given once a day. This dose is also effective and safe. Thus the dose to be provided in the GASTRANOX study is not markedly different from the high-risk doses already in routine clinical practice either in North America (30mg twice a day - 60mg total daily dosing) or 40mg once a day in Europe. It is also half of the full treatment dose which has been shown to be effective and safe in the treatment of venous thromboembolism.

Since cancer patients are recognised to have bleeding risk it was felt inappropriate to provide the full treatment dose of Enoxaparin. Thus half the full treatment doses provided. On the other hand the biological effect of low molecular weight heparins in cancer suggests that higher doses be given to enhance the potential survival benefit.

The study is intended to evaluate the safety and efficacy of the study drug compared to best normal practice. The standard methodology for such a comparison is to conduct a randomized, comparative study.

Multi-centre: It is anticipated that a single centre will be unable to recruit sufficient subjects, in 1 year, to conduct the assessment and therefore multiple centres will be recruited to conduct the study.

Open Label: All patients will receive standard care at their site. It would not be feasible to expect placebo parenteral administration for six months. All VTE events will be adjudicated. Mortality is an objective end-point.

Standard treatment control: subjects will be treated according to best practice with half also receiving the study treatment.

Parallel-group: due to the nature of the condition this is the only practical design.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or Female of age 18-75 years
* Histologically confirmed gastric or gastro-oesophageal carcinoma.
* Adenocarcinoma of the stomach stage III or IV considered inoperable at presentation.
* ECOG performance status ≤ 1
* Criteria for chemotherapy fulfilled (haematological, hepatic, renal).
* Ability to receive daily injection (self-injection or by patient relative).
* Urine-Pregnancy test negative.
* Consent to the use of Contraceptive for women of child bearing age group

Exclusion Criteria:

* History of previous malignancy within the previous 5 years (except curatively treated carcinoma in situ of the uterine cervix, or basal cell carcinoma of the skin), or concomitant malignancy.
* Prior treatment with chemotherapy or radiotherapy if relapse less than 6 months
* Non-epithelial gastric tumours, borderline tumours.
* Medically unstable patients, including but not limited to those with active infection, acute hepatitis, gastrointestinal bleeding, uncontrolled cardiac arrhythmias, interstitial lung disease, inflammatory bowel disease, uncontrolled angina, uncontrolled hypercalcaemia, uncompensated congestive heart failure, uncontrolled diabetes, persistent renal failure, dementia, seizures, superior vena cava syndrome.
* Persistent renal failure (persistent value of the calculated creatinine clearance < 30 mL/min defined as a documented value < 30 mL/min on at least 2 occasions ≥ 3 days prior entry into the study).
* Prosthetic heart valves.
* Any evidence of active bleeding disorder or risk of bleeding identified on fibroscopy done as a routine investigation before the consent for the trial. Fibroscopy is not mandatory to be done for the trial
* Current, objectively-verified DVT, PE or other clinically significant thrombosis.
* Documented previous episode of heparin-induced thrombocytopenia and/or thrombosis (HIT, HAT, or HITTS).
* Contraindications to anticoagulation
* Coagulopathies (acquired or inherited)
* Prior history of cerebral hemorrhage or neurosurgery within the previous month
* Bacterial endocarditis
* Uncontrolled arterial hypertension (systolic BP:200 mmHg or diastolic BP:110 mmHg) at 2 successive readings
* Haemostatic abnormalities: circulating anticoagulant, baseline platelet count <50 000/mm3, activated partial thromboplastin time (aPTT) value 1.5 x the upper limit of normal, or International Normalized Ratio (INR) >1.5. The laboratory test valid would be no earlier than 14 days for this criterion.
* Indication for thrombolytic therapy
* Any long-term anticoagulant therapy for medical condition.
* Immunocompromised subjects, such as subjects with known HIV and those who have either had an AIDS-defining condition (e.g. Kaposi's sarcoma, Pneumocystitis carinii pneumonia) or have CD4 + T-lymphocyte count < 200 /mm3.
* Known hypersensitivity to heparin, or LMWH, or pork derived products.
* Body weight >100 kg.
* Pregnant or lactating women.
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling to be tested for pregnancy (pregnancy status should be checked by serum or urine pregnancy testing prior to exposure to the investigational product
* Participation in another clinical trial (study medications / study devices) within the previous 30 days. (Surgical trials are allowed).
* Psychiatric disorders of altered mentation that would preclude understanding of the informed consent process.
* Psychological, familial, sociological, or geographical conditions, which do not permit treatment and/or medical follow-up required to comply with the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Event Free Survival (EFS) - Composite endpoint of overall survival plus free of symptomatic VTE . | up to 1 year from start of treatment

SECONDARY OUTCOMES:
Incidence of SVTE Overall survival Major and minor haemorrhages during chemotherapy and / or up to 30 days after last dose is provided. Serious adverse events, All reported adverse events HIT | upto 1 year from the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K Kakkar, PhD, Principal Investigator — Thrombosis Research Institute
Locations (15):
- India (15):
  - Mahatma Gandhi Cancer Hospital & Research Institute ,1/7 M.V.P. Colony, - ,, ., Vishakhapattanam, Andhra Pradesh
  - Mahavir Cancer Sansthan,Phulwari Sharif, Patna, Bihar
  - Gujarat Cancer Research Institute, Civil Hospital Campus,Asarwa, ,, Ahmedabad, Gujarat
  - Department Of Radiotherapy,S.S.G. Hospital, -, Baroda,Vadodara, Gujarat
  - Gokula Curie Cancer Centre,M.S.Ramaiah Memorial Hospital,MSR Nagar, MSRIT Post, Bangalore, Karnataka
  - Madhavan J.P., Trivandrum, Kerala
  - MGM Medical College & MY Hospital,, Indore, M.P
  - Cancer Hospital & Research Institute, Cancer Hill, Gwalior, Madhya Pradesh
  - Curie Manavta Cancer Centre, Opp.Hotel Sandeep Naka,Nashik, Mumbai, Maharashtra
  - Ruby Hall Clinic,Cancer Building,40 sassoon Road, , ,, Pune, Maharashtra
  - Acharya Tulsi Regional Cancer Treatment & Research Institute, Bikaner, Uttar Pradesh
  - B.P.Poddar Hospital & Medical Research Ltd,71/1, Humayun Kabir Sarani,, Block-G, New Alipore, Kolkata, West Bangol
  - Chittaranjan National Cancer Institute,37, S.P.Mukhurjee Road, Kolkata, West Bengal
  - Biswajit Sanyal, Kolkata, West Bengal
  - Dr. BRA IRCH,all India Institute of Medical Sciences,Ansari Nagar,, New Delhi

REFERENCES:
- [Background] Parkin DM, Bray FI, Devesa SS. Cancer burden in the year 2000. The global picture. Eur J Cancer. 2001 Oct;37 Suppl 8:S4-66. doi: 10.1016/s0959-8049(01)00267-2. No abstract available. PMID 11602373
- [Background] Lee YJ, Jy W, Horstman LL, Janania J, Reyes Y, Kelley RE, Ahn YS. Elevated platelet microparticles in transient ischemic attacks, lacunar infarcts, and multiinfarct dementias. Thromb Res. 1993 Nov 15;72(4):295-304. doi: 10.1016/0049-3848(93)90138-e. PMID 8303669
- [Background] Powell J, McConkey CC. The rising trend in oesophageal adenocarcinoma and gastric cardia. Eur J Cancer Prev. 1992 Apr;1(3):265-9. doi: 10.1097/00008469-199204000-00008. PMID 1467772
- [Background] Greenlee RT, Murray T, Bolden S, Wingo PA. Cancer statistics, 2000. CA Cancer J Clin. 2000 Jan-Feb;50(1):7-33. doi: 10.3322/canjclin.50.1.7. PMID 10735013
- [Background] Cohen AT, Wagner MB, Mohamed MS. Risk factors for bleeding in major abdominal surgery using heparin thromboprophylaxis. Am J Surg. 1997 Jul;174(1):1-5. doi: 10.1016/S0002-9610(97)00050-0. PMID 9240942
- [Background] Ajani JA. Chemotherapy for gastric carcinoma: new and old options. Oncology (Williston Park). 1998 Oct;12(10 Suppl 7):44-7. PMID 9830625
- [Background] Panzini I, Gianni L, Fattori PP, Tassinari D, Imola M, Fabbri P, Arcangeli V, Drudi G, Canuti D, Fochessati F, Ravaioli A. Adjuvant chemotherapy in gastric cancer: a meta-analysis of randomized trials and a comparison with previous meta-analyses. Tumori. 2002 Jan-Feb;88(1):21-7. PMID 12004845
- [Background] Petralia GA, Lemoine NR, Kakkar AK. Mechanisms of disease: the impact of antithrombotic therapy in cancer patients. Nat Clin Pract Oncol. 2005 Jul;2(7):356-63. doi: 10.1038/ncponc0225. PMID 16075795
- [Background] Thodiyil PA, Kakkar AK. Variation in relative risk of venous thromboembolism in different cancers. Thromb Haemost. 2002 Jun;87(6):1076-7. No abstract available. PMID 12083490
- [Background] Mismetti P, Laporte S, Darmon JY, Buchmuller A, Decousus H. Meta-analysis of low molecular weight heparin in the prevention of venous thromboembolism in general surgery. Br J Surg. 2001 Jul;88(7):913-30. doi: 10.1046/j.0007-1323.2001.01800.x. PMID 11442521
- [Background] Bergqvist D, Agnelli G, Cohen AT, Eldor A, Nilsson PE, Le Moigne-Amrani A, Dietrich-Neto F; ENOXACAN II Investigators. Duration of prophylaxis against venous thromboembolism with enoxaparin after surgery for cancer. N Engl J Med. 2002 Mar 28;346(13):975-80. doi: 10.1056/NEJMoa012385. PMID 11919306
- [Background] Rasmussen MS. Does prolonged thromboprophylaxis improve outcome in patients undergoing surgery? Cancer Treat Rev. 2003 Jun;29 Suppl 2:15-7. doi: 10.1016/s0305-7372(03)80004-x. PMID 12887945
- [Background] Kakkar AK, Levine MN, Kadziola Z, Lemoine NR, Low V, Patel HK, Rustin G, Thomas M, Quigley M, Williamson RC. Low molecular weight heparin, therapy with dalteparin, and survival in advanced cancer: the fragmin advanced malignancy outcome study (FAMOUS). J Clin Oncol. 2004 May 15;22(10):1944-8. doi: 10.1200/JCO.2004.10.002. PMID 15143088
- [Background] Altinbas M, Coskun HS, Er O, Ozkan M, Eser B, Unal A, Cetin M, Soyuer S. A randomized clinical trial of combination chemotherapy with and without low-molecular-weight heparin in small cell lung cancer. J Thromb Haemost. 2004 Aug;2(8):1266-71. doi: 10.1111/j.1538-7836.2004.00871.x. PMID 15304029
- [Background] Lee AY, Levine MN, Baker RI, Bowden C, Kakkar AK, Prins M, Rickles FR, Julian JA, Haley S, Kovacs MJ, Gent M; Randomized Comparison of Low-Molecular-Weight Heparin versus Oral Anticoagulant Therapy for the Prevention of Recurrent Venous Thromboembolism in Patients with Cancer (CLOT) Investigators. Low-molecular-weight heparin versus a coumarin for the prevention of recurrent venous thromboembolism in patients with cancer. N Engl J Med. 2003 Jul 10;349(2):146-53. doi: 10.1056/NEJMoa025313. PMID 12853587
- [Background] Klerk CPW SS, Otten JMM, Buller HR, on behalf of the MALT Stusy Group. Malignancy and low molwcular weight heparin therapy: the MALT trial. Phathophysiology of Haemostasis and Thrombosis 2003; 33(Suppl 1):75.
- [Background] von Tempelhoff GF, Harenberg J, Niemann F, Hommel G, Kirkpatrick CJ, Heilmann L. Effect of low molecular weight heparin (Certoparin) versus unfractionated heparin on cancer survival following breast and pelvic cancer surgery: A prospective randomized double-blind trial. Int J Oncol. 2000 Apr;16(4):815-24. doi: 10.3892/ijo.16.4.815. PMID 10717252
- [Background] Lee AY, Rickles FR, Julian JA, Gent M, Baker RI, Bowden C, Kakkar AK, Prins M, Levine MN. Randomized comparison of low molecular weight heparin and coumarin derivatives on the survival of patients with cancer and venous thromboembolism. J Clin Oncol. 2005 Apr 1;23(10):2123-9. doi: 10.1200/JCO.2005.03.133. Epub 2005 Feb 7. PMID 15699480